CLINICAL TRIAL: NCT06006572
Title: Direct Anterior Approach of the Hip and Variations in Wound Complications Using Different Closure Techniques
Brief Title: Hip DAA Closure Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CKRU2023-1674
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Total Hip Replacement; Wound Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive (Active Comparator): After surgery, the closure technique utilized by the surgeons will be wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive
  Interventions: Procedure: wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive
- wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive (Active Comparator): After surgery, the closure technique utilized by the surgeons will be wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive
  Interventions: Procedure: wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive

INTERVENTIONS:
Procedure: wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive — wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive
  Arms: wound closure subcuticular running stitch using 3-0 monocryl suture without skin adhesive
Procedure: wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive — wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive
  Arms: wound closure subcuticular running stitch using 3-0 monocryl suture with two layers of skin adhesive

SUMMARY:
This study aims to analyze the difference in rates of wound complications using two different closure techniques in Direct anterior approach for primary total hip replacement.

DETAILED DESCRIPTION:
The use of the direct anterior approach (DAA) for primary total hip arthroplasty (THA) has been increasingly popular but there has been a reported increased risk of wound complications compared with a posterior approach. Wound complications can lead to increased length of stay, reoperation procedures (i.e., irrigation and debridement), patient dissatisfaction, extra visits, readmissions, increased risk of periprosthetic joint infection and overall increased costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old that will undergo THA via DAA

Exclusion Criteria:

* Previous hip arthroplasty surgeries or scars
* THA secondary to oncologic or traumatic etiologies
* BMI ≥ 40
* uncontrolled diabetes (measured by a Hgb A1c above 8)
* reported allergy to skin adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Wound complications | 90 days
  Assessed using photographic documentation of the wound
Participant satisfaction | 90 days
  assessed using the POSAS (patient and observer scar assessment scale) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States